CLINICAL TRIAL: NCT00904969
Title: A Pre-Market Study of the AMS Transobturator Male Sling System for the Treatment of Male Stress Urinary Incontinence
Brief Title: A Pre-Market Study of the American Medical Systems (AMS) Transobturator Male Sling System for the Treatment of Male Stress Urinary Incontinence
Acronym: AMS051
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMS051
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2017-01

CONDITIONS: Urinary Incontinence, Stress
Keywords: Urinary Incontinence, Stress; Intrinsic sphincter deficiency; Secondary; Transurethral Resection (TUR); Transurethral Resection of the Prostate (TURP); Radical prostatectomy; Open prostatectomy; Post-suprapubic prostatectomy
MeSH Terms: conditions — Urinary Incontinence, Stress; Neoplasm Metastasis | interventions — Suburethral Slings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMS Transobturator Male Sling System (Experimental)
  Interventions: Device: The AMS Male Transobturator Sling System; Device: AdVance Male Sling

INTERVENTIONS:
Device: The AMS Male Transobturator Sling System — The AMS Male Transobturator Sling System was developed to treat urinary stress incontinence in men resulting from intrinsic sphincter deficiency (ISD) secondary to radical prostatectomy. The Male Transobturator Sling System procedure is minimally invasive and consists of using two single-use needle passers and passing them through two small incisions over the obturator foramen. The needles are pushed in an arc through the tissue and exited at a perineal incision. Once the passers are through the perineal incision, the Sling System mesh arms are attached to the needles which are then pulled back through the needle track to their points of origin over the obturator foramen. The Sling System is subsequently tensioned and all incisions are closed.
Device: AdVance Male Sling — A transobturator sling for the treatment of post-prostatectomy incontinence
  Other Names: Male TO; transobturator sling; suburethral sling; retrourethral sling

SUMMARY:
The purpose of this study is to obtain surgical technique data for use in physician education and training and to collect early clinical outcomes data for future publication.

DETAILED DESCRIPTION:
A multi-center study conducted under a common implant and follow-up protocol. The study will collect pre-operative urologic testing, medical history and subject quality of life (Incontinence Quality of Life Questionnaire). Intra-operative procedural data will be collected.

Pad weight and incontinence severity rating (using the International Consultation on Incontinence Questionnaire (ICIQ)) will be used to characterize continence status.

Post-operative complications, urologic testing, and subject quality of life will be collected at six weeks and three, six, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has agreed to be implanted with the AMS Male Transobturator Sling System.
2. The subject is willing and able to give valid informed consent.
3. The subject is > 40 years of age.
4. The subject has confirmed stress urinary incontinence for at least 6 months and uses no more than 8 pads per day for incontinence management.
5. The subject has any of the following: an observable degree of incontinence during stress related activities, more than one pad is used in a 24 hour period, has more than two episodes of incontinence per day.
6. Internal sphincter contractility confirmed by endoscopic view.
7. The subject's primary etiology is TUR, TURP, radical prostatectomy, open prostatectomy, or suprapubic prostatectomy
8. Pre-existing urological conditions, other than incontinence have been treated and are under control.
9. The subject is willing and able to return for follow-up evaluations and questionnaire completion according to the study protocol.
10. The subject is a good surgical candidate.

Exclusion Criteria:

1. The subject has a neurogenic bladder condition that is not treatable or controllable by pharmacological or alternative methods.
2. The subject has an atonic bladder.
3. The subject has a post-void residual > 75 cc.
4. The subject has detrusor-external sphincter dyssynergia.
5. The subject has a urinary tract infection (UTI).
6. The subject was treated with pelvic radiation within the last 6 months.
7. The subject currently has an inflatable penile prosthesis.
8. The subject self-catheterizes.
9. The subject has symptomatic or unstable bladder neck stricture disease.
10. The subject has a history of urethral strictures that may require repetitive instrumentation.
11. The subject has previously had a urethral Sling System, an AMS Sphincter 800™, or any implanted device for the treatment of urinary incontinence (not including bulking agents).
12. The subject has a history of connective tissue or autoimmune conditions.
13. The subject has a compromised immune system.
14. The subject has renal insufficiency, and upper and/or lower urinary tract relative obstruction.
15. The subject's reading level is judged inadequate for reading and understanding the quality of life questionnaires and other study materials.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-09; Primary Completion 2009-05 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Bales, M.D., Principal Investigator — University of Chicago Hospital; Timothy Boone, M.D., Principal Investigator — Baylor College of Medicine; Karyn Eilber, M.D., Principal Investigator — Century City Doctors Hospital; Brian J. Flynn, M.D., Principal Investigator — University of Colorado Health; Michael Guralnick, M.D., Principal Investigator — Medical College of Wisconsin; Sender Herschorn, M.D., Principal Investigator — Sunnybrook Health Sciences Centre; LeRoy Jones, M.D., Principal Investigator — CHRISTUS Health; Gerald Jordan, M.D., Principal Investigator — Norfolk General; Michael Kennelly, M.D., Principal Investigator — CHCS - Carolinas Medical Center; Dean L. Knoll, M.D., Principal Investigator — Centennial Hospital; Edward McGuire, M.D., Principal Investigator — The University of Michigan HS; Brian Roberts, M.D., Principal Investigator — Carolina Urologic Research Center; George D. Webster, M.D., Principal Investigator — Duke University
Locations (11):
- United States (10):
  - Century City Docotrs Hospital, Los Angeles, California
  - University of Colorado Health, Denver, Colorado
  - The University of Michigan HS, Ann Arbor, Michigan
  - CHCS - Carolinas Medical Center, Charlotte, North Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Centennial Hospital, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Christus Santa Rosa Hospital, San Antonio, Texas
  - Norfolk General, Norfolk, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data generated from this study may be used to support clinical publications, internal device documents for marketing and/or instructional manuals, etc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 clinical Sites enrolled and implanted subjects. All subjects gave informed consent prior to enrollment and all implanted subjects met the inclusion / exclusion criteria. Enrollment into the study began in February 2006 and ended April 2007.
Pre-assignment Details: Subjects who meet the inclusion / exclusion criteria and were good surgical candidates were enrolled into the single arm study and were eligible to be implanted.
Groups:
- Treated Participants: Participants in which a device placement was attempted.
Period: Overall Study
Arm/Group | Treated Participants
Started | 50 (Number of patients with an attempted implant; 1 subject with procedure aborted)
Completed | 31 (# of Implanted Subjects Who Completed the Study)
Not Completed | 19
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 3
Not completed — Additional Treatments | 11
Not completed — Case Aborted; Subject Exited | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 50
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 39
  African American | 10
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 48
  Canada | 2
Primary etiology of intrinsic sphincter deficiency (ISD) [Number; unit: participants]
  Post-Transurethral Resection of Prostate (TURP) | 3
  Radical Prostatectomy | 47
Years Since Surgery [Number; unit: participants]
  <=1995 | 7
  1996 - 2001 | 14
  2002-2004 | 18
  2005 | 8
  2006 | 3
Duration of Incontinence Symptoms [Mean (Standard Deviation); unit: months] | 57.2 (76.5)

OUTCOME MEASURES:

1. Primary Outcome: Procedural Endpoint: Procedure Time From First Incision to Closing.
Description: Characterize procedure time from first incision to closing.
Time Frame: During Procedure, Approximately 60 Minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
minutes | 61.8 (25.4)

2. Primary Outcome: Procedural Endpoint: Type of Anesthesia Used
Description: Describe the type of anesthesia used.
Time Frame: During Procedure, Approximately 60 Minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
Participants
  General | 41
  Spinal | 9

3. Primary Outcome: Procedural Endpoint: Rate of Foley Catheter Use - Intraoperative
Description: Number of participants requiring the use of a foley catheter intra-operatively.
Time Frame: During Procedure, Approximately 60 Minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
Participants | 44

4. Primary Outcome: Procedural Endpoint: Rate of Foley Catheter Use - Post-operative
Description: Number of participants requiring the use of a foley catheter who were able to void prior to discharge.
Time Frame: post-operative to discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
Participants | 39

5. Primary Outcome: Procedural Endpoint: Rate of Foley Catheter Use - Post-discharge
Description: Number of participants requiring the use of a foley catheter post-discharge following Bladder Management instructions.
Time Frame: post discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
Participants
  No instructions | 35
  Intermittent self-catheterization | 5
  Foley catheter | 10

6. Primary Outcome: Procedural Endpoint: Descriptive Procedural Parameters - Use of Tack Sutures
Description: Characterize procedural parameters including the use of tack sutures.
Time Frame: During Procedure, Approximately 60 Minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
Participants
  Tack suture used | 45
  Corpus spongiosum | 37
  Perineal body | 16
  Other tack suture | 9

7. Primary Outcome: Procedural Endpoint: Descriptive Procedural Parameters - Muscle Dissection
Description: Characterize procedural parameters, including muscle dissection across all participants.
Time Frame: During Procedure, Approximately 60 Minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
Participants | 50

8. Primary Outcome: Procedural Endpoint: Descriptive Procedural Parameters - Movement of Urethral Bulb While Tensioning
Description: Characterize procedural parameters, including the movement of urethral bulb while tensioning in all participants.
Time Frame: During Procedure, Approximately 60 Minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
Participants
  2 cm | 5
  3 cm | 34
  > 3 cm | 11

9. Primary Outcome: Device Success as Defined as Successful Placement of the Device in Desired Position Peri-operatively
Description: Summarize device success as defined as a successful placement of the device in a desired position, peri-operatively, in participants.
Time Frame: During Procedure, Approximately 60 Minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
Participants | 49

10. Secondary Outcome: Subject Satisfaction Endpoint: 1-Hour Pad Weight
Description: Summarize subject satisfaction of 1-hour pad weight for participants.
Time Frame: Baseline to 24 month
Population: Last observation carried forward (LOCF) and worst case scenario (WCS) data are derived from data from the 24 month visit
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
grams
  Baseline: number analyzed (Participants) | 48
  Baseline | 78.4 (102.3)
  3 Month: number analyzed (Participants) | 39
  3 Month | 8.9 (24.2)
  6 Month: number analyzed (Participants) | 37
  6 Month | 23.6 (49.5)
  12 Month: number analyzed (Participants) | 33
  12 Month | 15.8 (29.7)
  24 Month: number analyzed (Participants) | 39
  24 Month | 21.0 (67.0)
  24 Month LOCF: number analyzed (Participants) | 41
  24 Month LOCF | 22.2 (59.2)
  24 Month WCS: number analyzed (Participants) | 48
  24 Month WCS | 30.5 (76.1)

11. Secondary Outcome: Subject Satisfaction Endpoint: 24-Hour Pad Weight
Description: Summarize subject satisfaction with 24-hour pad weight across participants.
Time Frame: Baseline to 24 month
Population: LOCF and WCS data are derived from data from the 24 month visit
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
grams
  Baseline: number analyzed (Participants) | 48
  Baseline | 377.2 (657.5)
  3 Month: number analyzed (Participants) | 32
  3 Month | 108.0 (191.7)
  6 Month: number analyzed (Participants) | 30
  6 Month | 53.7 (99.1)
  12 Month: number analyzed (Participants) | 31
  12 Month | 42.0 (92.3)
  24 Month: number analyzed (Participants) | 28
  24 Month | 38.3 (58.8)
  24 Month LOCF: number analyzed (Participants) | 42
  24 Month LOCF | 73.0 (131.2)
  24 Month WCS: number analyzed (Participants) | 48
  24 Month WCS | 110.0 (244.1)

12. Secondary Outcome: Subject Satisfaction Endpoint: Percentage of Subjects Having a Decrease of Pad Weight of 25%, 50%, or 75% at Follow-Up. (1 Hour Pad Weight Test)
Description: Summarize the percent of subjects that have a decrease of pad weight of 25%, 50%, or 75% at follow-up (1-hour pad weight test used).
Time Frame: Baseline to 24 month
Measure: Number; unit: participants
Groups:
- 3 Month: 3 Month Follow-Up Visit
- 6 Month: 6 Month Follow-Up Visit
- 12 Month: 12 Month Follow-Up Visit
- 24 Month: 24 Month Follow-Up Visit
- 24 Month LOCF: 24 Month Visit using Last Observation Carried Forward
- 24 Month WCS: 24 Month Visit using Worse Case Scenario
Arm/Group | 3 Month | 6 Month | 12 Month | 24 Month | 24 Month LOCF | 24 Month WCS
Number analyzed (Participants) | 39 | 37 | 33 | 29 | 41 | 48
participants
  1-Hour ≥ 25% Reduction in Pad Weight | 34 | 28 | 29 | 25 | 34 | 34
  1-Hour ≥ 50% Reduction in Pad Weight | 32 | 25 | 25 | 24 | 31 | 31
  1-Hour ≥ 75% Reduction in Pad Weight | 26 | 24 | 23 | 20 | 26 | 26

13. Secondary Outcome: Subject Satisfaction Endpoint: Percentage of Subjects Having a Decrease of Pad Weight of 25%, 50%, or 75% at Follow-Up. (24 Hour Pad Weight Test)
Description: Summarize the percent of subjects that have a decrease of pad weight of 25%, 50%, or 75% at follow-up (24-hour pad weight test used).
Time Frame: Baseline to 24 Month
Measure: Number; unit: participants
Arm/Group | 3 Month | 6 Month | 12 Month | 24 Month | 24 Month LOCF | 24 Month WCS
Number analyzed (Participants) | 32 | 30 | 31 | 28 | 42 | 48
participants
  24-Hour ≥ 25% Reduction in Pad Weight | 26 | 28 | 29 | 26 | 36 | 36
  24-Hour ≥ 50% Reduction in Pad Weight | 24 | 24 | 27 | 26 | 34 | 34
  24-Hour ≥ 75% Reduction in Pad Weight | 20 | 22 | 25 | 20 | 26 | 26

14. Secondary Outcome: Subject Satisfaction Endpoint: Pads Per Day Use
Description: Summarize the subject satisfaction using pads per day use collected in follow-up in participants.
Time Frame: Baseline to 24 Months
Population: LOCF and WCS data are derived from data from the 24 month visit
Measure: Count of Participants; unit: Participants
Groups:
- 0-1 PPD: 0-1 Pads per Day Use
- 2-3 PPD: 2-3 Pads per Day Use
- 4-5 PPD: 4-5 Pads per Day Use
- 6-7 PPD: 6-7 Pads per Day Use
- >= 10 PPD: Greater than or equal to 10 Pads per Day Use
Arm/Group | 0-1 PPD | 2-3 PPD | 4-5 PPD | 6-7 PPD | >= 10 PPD
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50
Participants
  Baseline: number analyzed (Participants) | 49 | 49 | 49 | 49 | 49
  Baseline | 7 | 20 | 13 | 8 | 1
  6 Week: number analyzed (Participants) | 48 | 48 | 48 | 48 | 48
  6 Week | 33 | 8 | 2 | 2 | 3
  3 Month: number analyzed (Participants) | 44 | 44 | 44 | 44 | 44
  3 Month | 34 | 6 | 2 | 2 | 0
  6 Month: number analyzed (Participants) | 39 | 39 | 39 | 39 | 39
  6 Month | 32 | 4 | 3 | 0 | 0
  12 Month: number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
  12 Month | 26 | 7 | 2 | 1 | 1
  24 Month: number analyzed (Participants) | 31 | 31 | 31 | 31 | 31
  24 Month | 21 | 9 | 1 | 0 | 0
  24 Month LOCF: number analyzed (Participants) | 49 | 49 | 49 | 49 | 49
  24 Month LOCF | 25 | 15 | 3 | 3 | 3
  24 Month WCS: number analyzed (Participants) | 49 | 49 | 49 | 49 | 49
  24 Month WCS | 25 | 15 | 3 | 3 | 3

15. Secondary Outcome: Subject Satisfaction Endpoint: Quality of Life I-QOL Scores
Description: The Incontinence Quality of Life (I-QOL) questionnaire contains 22 items, each with a 5-point Likert-type response scale, evaluating a subject's quality of life with respect to his urinary problems or incontinence. A possible total score can be 0-100, with a higher score meaning less problems.
Time Frame: Baseline to 24 Months
Population: Number of subjects that did not have test performed at follow-up visit.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
score
  Baseline: number analyzed (Participants) | 49
  Baseline | 50.3 (22.4)
  3 Month: number analyzed (Participants) | 40
  3 Month | 79.2 (20.9)
  6 Month: number analyzed (Participants) | 39
  6 Month | 79.4 (21.6)
  12 Month: number analyzed (Participants) | 35
  12 Month | 79.9 (22.9)
  24 Month: number analyzed (Participants) | 31
  24 Month | 82.4 (18.3)

16. Secondary Outcome: Subject Satisfaction Endpoint: Quality of Life International Consultation on Incontinence Questionnaire Short-Form (ICIQ-SF) Scores
Description: The ICIQ-SF questionnaire evaluates the impact of urinary incontinence on quality of life through four questions that evaluate the frequency, severity and impact of urinary incontinence. A set of eight self-diagnosis items related to the causes or situations of urinary incontinence experienced by the subject are also assessed. Scores may range from 0 to 21. Improvement in the subject's quality of life from baseline to follow-up is indicated by a decrease in the ICIQ-SF score.
Time Frame: Baseline to 24 Months
Population: Number of subjects that did not have test performed at follow-up visit.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
score
  Baseline: number analyzed (Participants) | 49
  Baseline | 15.7 (4.1)
  3 Month: number analyzed (Participants) | 41
  3 Month | 7.6 (5.6)
  6 Month: number analyzed (Participants) | 39
  6 Month | 7.6 (5.7)
  12 Month: number analyzed (Participants) | 35
  12 Month | 7.3 (5.8)
  24 Month: number analyzed (Participants) | 31
  24 Month | 7.5 (5.5)

17. Post Hoc Outcome: Uroflow Studies: Peak Flow Rate
Description: Baseline uroflow measurements including peak flow rates, average flow rates, voided volume, and post-void residual were compared to follow-up results at 3, 6, 12, and 24 months.
Time Frame: Baseline to 24 month
Population: Number of subjects that did not have test performed at follow-up visit.
Measure: Mean (Standard Deviation); unit: ml/sec
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
ml/sec
  Baseline: number analyzed (Participants) | 49
  Baseline | 20.8 (11.3)
  3 Month: number analyzed (Participants) | 38
  3 Month | 20.9 (13.5)
  6 Month: number analyzed (Participants) | 37
  6 Month | 19.8 (13.8)
  12 Month: number analyzed (Participants) | 35
  12 Month | 19.4 (8.4)
  24 Month: number analyzed (Participants) | 28
  24 Month | 20.1 (8.5)

18. Post Hoc Outcome: Uroflow Studies: Average Flow Rates
Description: as for outcome 17
Time Frame: Baseline to 24 Month
Population: Number of subjects that did not have test performed at follow-up visit.
Measure: Mean (Standard Deviation); unit: ml/sec
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
ml/sec
  Baseline: number analyzed (Participants) | 44
  Baseline | 12.0 (6.0)
  3 Month: number analyzed (Participants) | 38
  3 Month | 11.1 (7.0)
  6 Month: number analyzed (Participants) | 36
  6 Month | 11.3 (9.8)
  12 Month: number analyzed (Participants) | 35
  12 Month | 10.9 (4.9)
  24 Month: number analyzed (Participants) | 28
  24 Month | 11.5 (5.8)

19. Post Hoc Outcome: Uroflow Studies: Voided Volume
Description: as for outcome 17
Time Frame: Baseline to 24 Months
Population: Number of subjects that did not have test performed at follow-up visit.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
ml
  Baseline: number analyzed (Participants) | 49
  Baseline | 280.8 (112.4)
  3 Month: number analyzed (Participants) | 38
  3 Month | 263.0 (142.6)
  6 Month: number analyzed (Participants) | 37
  6 Month | 244.2 (114.3)
  12 Month: number analyzed (Participants) | 35
  12 Month | 248.7 (134.4)
  24 Month: number analyzed (Participants) | 28
  24 Month | 298.6 (147.4)

20. Post Hoc Outcome: Uroflow Studies: Post-Void Residual
Description: as for outcome 17
Time Frame: Baseline to 24 Months
Population: Number of subjects that did not have test performed at follow-up visit.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
ml
  Baseline: number analyzed (Participants) | 48
  Baseline | 17.0 (27.8)
  3 Month: number analyzed (Participants) | 39
  3 Month | 17.7 (31.1)
  6 Month: number analyzed (Participants) | 37
  6 Month | 23.8 (41.7)
  12 Month: number analyzed (Participants) | 35
  12 Month | 13.1 (30.0)
  24 Month: number analyzed (Participants) | 27
  24 Month | 18.2 (28.8)

21. Post Hoc Outcome: Urodynamic Results: Bladder Capacity
Description: Baseline urodynamic measurements including bladder capacity, maximum detrusor pressure, detrusor pressure at maximum flow, and detrusor instability were measured at baseline and at 6-month follow-up.
Time Frame: Baseline and 6 Months Post implant
Population: Number of subjects that did not have test performed at follow-up visit.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
ml
  Baseline: number analyzed (Participants) | 49
  Baseline | 323.5 (130.8)
  6 Month: number analyzed (Participants) | 34
  6 Month | 349.4 (136.7)

22. Post Hoc Outcome: Urodynamics Results: Maximum Detrusor Pressure
Description: Baseline urodynamic measurements including bladder capacity, maximum detrusor pressure, detrusor pressure at maximum flow, and detrusor instability were measured at baseline and at 6-month follow-up.
  Maximum detrusor pressure is measured during a urodynamic study when tension is applied to the bladder wall (detrusor muscles) by filling the bladder to capacity with saline water and observing the detrusor muscle during filling of the bladder and voiding of the saline water.
Time Frame: Baseline and 6 Months Post Implant
Population: Number of subjects that did not have test performed at follow-up visit.
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
cm H2O
  Baseline: number analyzed (Participants) | 46
  Baseline | 35.9 (27.4)
  6 Months: number analyzed (Participants) | 32
  6 Months | 32.3 (21.3)

23. Post Hoc Outcome: Urodynamics Results: Pdet at Qmax
Description: Baseline urodynamic measurements including bladder capacity, maximum detrusor pressure, detrusor pressure at maximum flow, and detrusor instability were measured at baseline and at 6-month follow-up.
  Maximum detrusor pressure is measured during a urodynamic study when tension is applied to the bladder wall (detrusor muscles) by filling the bladder to capacity with saline water and observing the detrusor muscle during filling of the bladder and voiding of the saline water. Pdet at Qmax is the detrusor pressure at maximal flow rate when the bladder is full and the patient begins voiding.
Time Frame: Baseline and 6 Months Post Implant
Population: Number of subjects that did not have test performed at follow-up visit.
Measure: Mean (Standard Deviation); unit: cm H20
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
cm H20
  Baseline: number analyzed (Participants) | 49
  Baseline | 26.2 (19.3)
  6 Months: number analyzed (Participants) | 32
  6 Months | 30.2 (17.1)

24. Post Hoc Outcome: Urodynamics Results: Detrusor Instability, Started at Filling Volume
Description: Baseline urodynamic measurements including bladder capacity, maximum detrusor pressure, detrusor pressure at maximum flow, and detrusor instability were measured at baseline and at 6-month follow-up.
  Detrusor instability occurs when the detrusor muscle is unstable and spontaneously contracts the bladder.
  The measure data table shows the mean volume at the start of the urodynamic measurement study for patients with detrusor instability.
Time Frame: Baseline and 6 Months Post Implant
Population: Number of subjects that did not have test performed at follow-up visit.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
ml
  Baseline: number analyzed (Participants) | 11
  Baseline | 225.8 (159.9)
  6 Month: number analyzed (Participants) | 4
  6 Month | 170.8 (32.1)

25. Post Hoc Outcome: Urodynamics Results: Detrusor Instability, Max Pdet
Description: Baseline urodynamic measurements including bladder capacity, maximum detrusor pressure, detrusor pressure at maximum flow, and detrusor instability were measured at baseline and at 6-month follow-up.
  Maximum detrusor pressure is measured during a urodynamic study when tension is applied to the bladder wall (detrusor muscles) by filling the bladder to capacity with saline water and observing the detrusor muscle during filling of the bladder and voiding of the saline water. Pdet at Qmax is the detrusor pressure at maximal flow rate when the bladder is full and the patient begins voiding.
  Detrusor instability occurs when the detrusor muscle is unstable and spontaneously contracts the bladder.
  The outcome measure data table shows the Pdet for patients with detrusor instability.
Time Frame: Baseline and 6 Months Post Implant
Population: Number of subjects that did not have test performed at follow-up visit.
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
cm H2O
  Baseline: number analyzed (Participants) | 11
  Baseline | 31.5 (31.3)
  6 Month: number analyzed (Participants) | 4
  6 Month | 41.0 (37.8)

26. Post Hoc Outcome: Urodynamics Results: Abnormal Cystometrogram, Abnormal End Fill Pressure
Description: Baseline urodynamic measurements including bladder capacity, maximum detrusor pressure, detrusor pressure at maximum flow, and detrusor instability were measured at baseline and at 6-month follow-up.
  Abnormal graphical representation of bladder pressure during urodynamics testing which is when the bladder is filled with saline water.
Time Frame: Baseline and 6 Months Post Implant
Population: Number of subjects that did not have test performed at follow-up visit.
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
cm H2O
  Baseline: number analyzed (Participants) | 7
  Baseline | 10.0 (8.3)
  6 Month: number analyzed (Participants) | 1
  6 Month | 6.0 (0)

27. Post Hoc Outcome: Urodynamic Results: Abdominal Leak Point Pressure
Description: Abdominal leak point pressure (ALPP) is one indicator of improvement in continence symptoms. Abdominal leak point pressure was collected at baseline and 6-month follow-up as part of the urodynamic assessment.
Time Frame: Baseline and 6 Months Post Implant
Population: 18 participants did not have 6-month follow-up data
Measure: Number; unit: participants
Arm/Group | Treated Participants
Number analyzed (Participants) | 31
participants
  Improved: leaked @ baseline, improved @ 6 months | 10
  Improved: leaked @ baseline, no leak @ 6 months | 14
  Unchanged: leaked same at baseline and 6 months | 1
  Unchanged: no leak @ baseline, no leak @ 6 months | 1
  Worsened: leaked @ baseline, leaked more at 6 mo | 4
  Worsened: no leak @ baseline, leak @ 6 months | 1

28. Secondary Outcome: Subject Satisfaction Endpoint: Quality of Life UCLA (University of California Los Angeles) / RAND (RAND Corporation) Scores
Description: Improvement in the subject's quality of life from baseline to follow-up is indicated by an increase in the UCLA/RAND urinary function score. Scores may range from 0 to 100.
Time Frame: Baseline to 24 Months
Population: Number of subjects that did not have test performed at follow-up visit.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
score
  Baseline: number analyzed (Participants) | 49
  Baseline | 20.1 (14.3)
  3 Month: number analyzed (Participants) | 41
  3 Month | 54.7 (28.7)
  6 Month: number analyzed (Participants) | 39
  6 Month | 55.9 (28.8)
  12 Month: number analyzed (Participants) | 35
  12 Month | 57.4 (29.1)
  24 Month: number analyzed (Participants) | 31
  24 Month | 57.3 (27.1)

29. Secondary Outcome: Subject Satisfaction Endpoint: Physician Evaluation of Subject's Incontinence Status
Description: Physician evaluation of subject's incontinence status at 6 weeks and subsequent follow-up evaluations
Time Frame: 6 Weeks post implant to 24 Months
Measure: Count of Participants; unit: Participants
Groups:
- Completely Dry: Defined as "No leakage".
- Substantially Improved: Defined as "May have periodic leakage of small amounts but additional protection not needed".
- Some Additional Protection May be Required: Defined as "Up to three pads per day may be needed or may wet themselves not more than once weekly".
- Substantially or Totally Incontinent: Defined as "Will require more than three pads per day or may wet themselves two or more times per week".
Arm/Group | Completely Dry | Substantially Improved | Some Additional Protection May be Required | Substantially or Totally Incontinent
Number analyzed (Participants) | 50 | 50 | 50 | 50
Participants
  6 Week | 12 | 17 | 12 | 7
  3 Month | 12 | 14 | 15 | 3
  6 Month | 12 | 11 | 14 | 2
  12 Month | 9 | 15 | 9 | 4
  24 Month | 7 | 12 | 11 | 1

30. Secondary Outcome: Procedural and Device Complication Rates
Description: Percentage of participants with serious and non-serious adverse events.
Time Frame: Procedure to 24 Months Post implant
Measure: Number; unit: percentage of participants
Arm/Group | Treated Participants
Number analyzed (Participants) | 50
percentage of participants | 54

ADVERSE EVENTS:
Time Frame: Adverse events were collected at the implant, 6 weeks, 3 month, 6 month, 12 month, and 24 month visits.
Description: Only adverse events related to the study device or procedure are displayed.
Arm/Group | Treated Participants
Serious Adverse Events (participants affected / at risk) | 2/50
Other Adverse Events (participants affected / at risk) | 25/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Participants (N=50)
Urinary Incontinence - Persistant (Renal and urinary disorders) | 1 (1)
Intra-operative Bleeding of Aberrant Vessel (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Participants (N=50)
Pain/ Discomfort (General disorders) | 8 (11)
Urinary retention (Renal and urinary disorders) | 10 (10)
Urinary Incontinence - Persistent (Renal and urinary disorders) | 3 (3)
Urinary Urgency (Renal and urinary disorders) | 2 (2)
Ecchymosis (Injury, poisoning and procedural complications) | 2 (2)
Post-Void Dribbling (Renal and urinary disorders) | 2 (2)
Pain/ Discomfort With Erections (Reproductive system and breast disorders) | 1 (1)
Urinary Incontinence - De Novo Stress (Renal and urinary disorders) | 1 (1)
Scrotal Pain/ Swelling (Injury, poisoning and procedural complications) | 1 (1)
Groin Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Decreased Penile Sensitivity (Nervous system disorders) | 1 (1)
Edema of Penis (Injury, poisoning and procedural complications) | 1 (1)
Light Post-Op Bleed (Injury, poisoning and procedural complications) | 1 (1)
Penile Pain with Orgasm (Reproductive system and breast disorders) | 1 (1)
Worsening Incontinence (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No